CLINICAL TRIAL: NCT03327324
Title: Improving Sleep Using Mentored Behavioral and Environmental Restructuring
Acronym: SLUMBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-00338; 1R01NR016461-01A1 (NIH)
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- F1U1 (Experimental): Sequence 1 (Facility 1/Unit 1): Baseline, then 3 Month SLUMBER Intervention, then 39 Month Sustainability.
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring
- F1U2 (Experimental): Sequence 2 (Facility 1/Unit 2): Baseline, then 3 Month SLUMBER Intervention, then 33 Month Sustainability
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring
- F2U2 (Experimental): Sequence 3 (Facility 2/Unit 2): Baseline, then 3 Month SLUMBER Intervention, then 27 Month Sustainability
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring
- F2U3 (Experimental): Sequence 4 (Facility 2/Unit 3): Baseline, then 3 Month SLUMBER Intervention, then 21 Month Sustainability
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring
- F2U4 (Experimental): Sequence 5 (Facility 2/Unit 4): Baseline, then 3 Month SLUMBER Intervention, then 15 Month Sustainability
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring
- F3U1 (Experimental): Sequence 6 (Facility 3/Unit 1): Baseline, then 3 Month SLUMBER Intervention, then 9 Month Sustainability
  Interventions: Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring

INTERVENTIONS:
Behavioral: Sleep Using Mentored Behavioral and Environmental Restructuring — SLUMBER is a non-pharmacological intervention program, delivered by providing mentoring to facility staff who work directly with residents. SLUMBER focuses on detecting sleep-disruptive factors including: nighttime noise and patient behaviors associated with poor sleep quality; disruptions caused by nighttime caregiving; daytime inactivity; and limited light exposure. In this model, staff-delivered interventions to improve these factors improve sleep quality thereby creating opportunities to test the impact of improving sleep quality (measured by actigraphy) on mood (depression and anxiety), pain, cognitive function, functional ability, and observed activity levels.
  Other Names: SLUMBER

SUMMARY:
The goal of this study is to test potential functional/psychosocial benefits of improved sleep using a program designed to teach nursing facility staff to improve sleep promoting strategies and environment for nursing home residents. Sleep disturbances are quite common in skilled nursing facilities and affect as many as 69% of residents while staff do not fully understand how to improve sleep without using medications. Medications for sleep are commonly used as first-line therapy for older adults but this is problematic because these medications can lead to greater problems with thinking, more frequent falls, and even worse sleep over time. In addition, poor sleep can lead to depressed mood, greater trouble with thinking and memory, worse pain, and greater need for help with daily activities.

DETAILED DESCRIPTION:
This is a study to test the effects of improved sleep quality on downstream functional/psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* living in the unit of intervention,
* ability to communicate and follow simple commands,
* English- or Spanish-speaking,
* capacity to consent assessed with standard questions used to assess capacity or having a surrogate who can provide consent.

Exclusion Criteria:

* Does not have capacity and does not show enthusiasm for the research
* Does not have capacity and does not have a proxy.
* obtunded or comatose state,
* inability to communicate verbally,
* inability to consent and without surrogate
* non-English and non-Spanish speaking. In keeping with QI strategies, all residents will be exposed to the environmental aspects of the intervention, as these strategies represent clinically proven non-experimental behavioral strategies with no perceptible harm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Chodosh J, Mitchell MN, Cadogan M, Brody AA, Alessi CA, Hernandez DE, Mangold M, Martin JL. Improving sleep using mentored behavioral and environmental restructuring (SLUMBER): A randomized stepped-wedge design trial to evaluate a comprehensive sleep intervention in skilled nursing facilities. Contemp Clin Trials. 2023 Mar;126:107107. doi: 10.1016/j.cct.2023.107107. Epub 2023 Jan 27. PMID 36716989

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a stepped wedge intervention trial (SWT). In this SWT, all units receive the intervention but at different time points. Every unit provides baseline and follow-up data.
Period: Baseline (Month 0-Month 3)
Arm/Group | F1U1 | F1U2 | F2U2 | F2U3 | F2U4 | F3U1
Started | 18 | 20 | 9 | 10 | 15 | 20
Completed | 18 | 17 | 9 | 9 | 13 | 14
Not Completed | 0 | 3 | 0 | 1 | 2 | 6
Not completed — Incomplete (participant did not complete all data items collected during study visit) | 0 | 1 | 0 | 1 | 0 | 5
Not completed — Refused | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — COVID-Incomplete (couldn't collect all subject data due to Nursing Home COVID shutdown) | 0 | 0 | 0 | 0 | 0 | 1
Period: Intervention (Month 3-Month 6)
Arm/Group | F1U1 | F1U2 | F2U2 | F2U3 | F2U4 | F3U1
Started | 18 | 17 | 9 | 9 | 13 | 14
Completed | 13 | 16 | 6 | 8 | 11 | 0
Not Completed | 5 | 1 | 3 | 1 | 2 | 14
Not completed — Incomplete (participant did not complete all data items collected during study visit) | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 1 | 0
Not completed — Left Nursing Home Facility | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 1 | 1 | 0
Not completed — COVID-Incomplete (couldn't collect all subject data due to Nursing Home COVID shutdown) | 0 | 0 | 0 | 0 | 0 | 14
Period: Sustainability Follow-Up 1 (Month 6-9)
Arm/Group | F1U1 | F1U2 | F2U2 | F2U3 | F2U4 | F3U1
Started | 13 | 16 | 6 | 8 | 11 | 0
Completed | 9 | 14 | 5 | 5 | 6 | 0
Not Completed | 4 | 2 | 1 | 3 | 5 | 0
Not completed — Incomplete (participant did not complete all data items collected during study visit) | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Left Nursing Home Facility | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0 | 0
Not completed — COVID-Incomplete (couldn't collect all subject data due to Nursing Home COVID shutdown) | 0 | 0 | 0 | 3 | 5 | 0
Period: Sustainability Follow-Up 2 (Month 9-12)
Arm/Group | F1U1 | F1U2 | F2U2 | F2U3 | F2U4 | F3U1
Started | 9 | 14 | 2 | 0 | 0 | 0
Completed | 7 | 14 | 2 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Left Nursing Home | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- F1U2: Sequence 2: (Facility 1/Unit 2): Baseline, then 3 Month SLUMBER Intervention, then 33 Month Sustainability
- Total: Total of all reporting groups
Arm/Group | F1U1 | F1U2 | F2U2 | F2U3 | F2U4 | F3U1 | Total
Number analyzed (Participants) | 18 | 17 | 9 | 9 | 13 | 14 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 66 (8) | 89 (7) | 92 (8) | 91 (5) | 75 (11) | 81 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 4 | 8 | 9 | 11 | 52
  Male | 9 | 6 | 5 | 1 | 4 | 3 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 2 | 0 | 2 | 2 | 17
  Not Hispanic or Latino | 13 | 11 | 7 | 9 | 11 | 12 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 9 | 0 | 0 | 1 | 3 | 26
  White | 0 | 2 | 7 | 7 | 10 | 9 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 2 | 0 | 2 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 9 | 9 | 13 | 14 | 80

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency (SE)
Description: Sleep efficiency (SE), commonly defined as the ratio of total sleep time (TST) to time in bed (TIB), will be reported as a percentage of time in bed. This data will be obtained from actigraphy analysis.
Time Frame: Baseline
Population: Sleep/wake time was measured using wrist actigraphs and some participants took off the watch, meaning some participants were not included in the analysis of this outcome measure.
Measure: Mean (95% Confidence Interval); unit: percentage of time in bed
Groups:
- Resident of the Skilled Nursing Facility: Sleep Using Mentored Behavioral and Environmental Restructuring: SLUMBER is a non-pharmacological intervention program, delivered by providing mentoring to facility staff who work directly with residents. SLUMBER focuses on detecting sleep-disruptive factors including: nighttime noise and patient behaviors associated with poor sleep quality; disruptions caused by nighttime caregiving; daytime inactivity; and limited light exposure. In this model, staff-delivered interventions to improve these factors improve sleep quality thereby creating opportunities to test the impact of improving sleep quality (measured by actigraphy) on mood (depression and anxiety), pain, cognitive function, functional ability, and observed activity levels.
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
percentage of time in bed | 76.1 [71.83 to 80.38]

2. Primary Outcome: Sleep Efficiency (SE)
Description: as for outcome 1
Time Frame: Post-Treatment (Month 6 Post-Baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of time in bed
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
percentage of time in bed | 75.69 [70.89 to 80.49]

3. Primary Outcome: Sleep Efficiency (SE)
Description: as for outcome 1
Time Frame: Month 9 Post-Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of time in bed
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
percentage of time in bed | 75.61 [70.05 to 81.18]

4. Primary Outcome: Nighttime Total Awake Time
Description: Data will be obtained from antigraphy analysis.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 11.54 [9.92 to 13.15]

5. Primary Outcome: Nighttime Total Awake Time
Description: Data will be obtained from antigraphy analysis.
Time Frame: Post-Treatment (Month 6 Post-Baseline)
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 11.03 [9.22 to 12.84]

6. Primary Outcome: Nighttime Total Awake Time
Description: Data will be obtained from antigraphy analysis.
Time Frame: Month 9 Post-Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 11.8 [9.29 to 14.31]

7. Primary Outcome: Daytime Sleeping (Napping) Time
Description: Wrist device / actigraphy will be used to measure sleep/wake time.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 305.91 [261.63 to 350.18]

8. Primary Outcome: Daytime Sleeping (Napping) Time
Description: Wrist device / actigraphy will be used to measure sleep/wake time.
Time Frame: Post-Treatment (Month 6 Post-Baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 369.7 [314.92 to 424.47]

9. Primary Outcome: Daytime Sleeping (Napping) Time
Description: Wrist device / actigraphy will be used to measure sleep/wake time.
Time Frame: Month 9 Post-Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 52
Minutes | 338.26 [287.79 to 388.73]

10. Primary Outcome: Score on Pittsburgh Sleep Quality Index (PSQI)
Description: PSQI contains 19 self-rated questions. The 19 questions are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The total score range is 0-21; the higher the score, the greater the difficulties in all areas.
Time Frame: Month 9 Post-Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 56
score on a scale | 6.5 [5.54 to 7.52]

11. Primary Outcome: Brief Anxiety and Depression Scale (BADS) Questionnaire Score
Description: BADS is a brief screening tool for mood impairment developed for older adults. It consists of 8 questions, answered 0 (no), 1(somewhat), or 2 (yes). The total score range is 0-16; the higher the score, the higher the level of mood impairment
Time Frame: Month 9 Post-Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 56
score on a scale | 5.15 [3.74 to 6.55]

12. Primary Outcome: Score on Brief Cognitive Assessment Tool (BCAT)
Description: BCAT is a multi-domain cognitive instrument that assesses orientation, verbal recall, visual recognition, visual recall, attention, abstraction, language, executive functions, and visuo-spatial processing in adult and older adult populations. It consists of 21 items. The total score range is 0-50; the higher the score, the more normal the level of cognitive functioning and independent living.
Time Frame: Month 9 Post-Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Resident of the Skilled Nursing Facility
Number analyzed (Participants) | 56
score on a scale | 28.33 [25.42 to 31.23]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Resident of the Skilled Nursing Facility
All-Cause Mortality (participants affected / at risk) | 9/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03327324/Prot_SAP_000.pdf